CLINICAL TRIAL: NCT03454399
Title: Does Transesophageal Echocardiography Along With an Orogastric Tube Improve the Image Quality Intraoperatively?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Yoshihisa Morita, Assistant professor, Henry Ford Health System
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 11078
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: TEE Image Quality

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEE image before suction (No Intervention): Suction orogastric tube which is attached to TEE probe
- TEE image after suction (Experimental): Suction orogastric tube which is attached to TEE probe
  Interventions: Procedure: Suction orogastric tube which is attached to TEE probe

INTERVENTIONS:
Procedure: Suction orogastric tube which is attached to TEE probe — Suction orogastric tube which is attached to TEE probe
  Arms: TEE image after suction

SUMMARY:
Image quality of intraoperative transesophageal echocardiography (TEE) tends to get worse during long hours of operations. An orogastric tube (OGT) is often inserted in the beginning of the case, and left there for intermittent suction as needed, or removed before TEE exam to prevent echoic artifacts. However, if left there, the effect of suction might be limited due to unreliable tip position of the OG tube. If removed, stomach will be distended again. We devised the OG tube attached TEE for practical suction and assessed its effect on image quality intraoperatively.

DETAILED DESCRIPTION:
OGT attached TEE probe is used for cardiac and liver transplantation cases. Each case is assigned 3 investigators who are blinded to this study design, We do image quality assessment by two methods; firstly, we categorize image quality as numbers based on each investigator's impression (1: Very bad, 2: bad, 3: acceptable, 4: good, 5: very good) and compare the difference in number before and after suctioning. Secondly, we evaluate consistency intraclass correlation coefficient (ICC) for inter-observer variability using investigator A, B and C. We evaluate absolute-agreement ICC for intra-observer variability using investigator C, who perform analysis for all images twice with a 6 to 8 months interval. This analysis was performed with left ventricular fraction area change using transgastric left ventricular short axis view.

ELIGIBILITY:
Inclusion Criteria:

* adult cardiac surgery or liver transplant surgery

Exclusion Criteria:

* TEE with significant wall motion abnormality or TEE contraindicated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Penning, MD, Study Director — HFHS
Locations (1):
- HFHS, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: image sets
Groups:
- TEE Image Before and After Suctioning Orogastric Tube: For intraoperative TEE used cardiac or liver transplant cases. TEE images will be stored before and after suctioning orogastric tube which is attached to TEE probe
Period: TEE Image Before Suction
Arm/Group | TEE Image Before and After Suctioning Orogastric Tube
Started | 47; 141 image sets
Completed | 47; 141 image sets
Not Completed | 0; 0 image sets
Period: TEE Image After Suction
Arm/Group | TEE Image Before and After Suctioning Orogastric Tube
Started | 47; 141 image sets
Completed | 47; 141 image sets
Not Completed | 0; 0 image sets

BASELINE CHARACTERISTICS:
Population: Surgeries which need intraoperative TEE
Groups:
- TEE Image Before and After Suction: Surgeries which need intraoperative TEE (i.e. cardiac surgery and orthotopic liver transplant)
Arm/Group | TEE Image Before and After Suction
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 7
Age, Continuous [Median (Standard Deviation); unit: years] | 62.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Image Quality Assessment Method#1: Difference in Likert Scale Before and After Suctioning
Description: Difference in image quality assessment by Likert scale before/after suctioning, by assessing quality of images stored before/after suctioning. Investigators categorized the quality of all acquired images on a numeric scale (the higher number means higher image quality) based on each investigator's impression (1: very poor, 2: poor, 3: acceptable, 4: good, and 5: very good). Image quality improvement was determined by increased number. Three investigators (A, B, C) assessed the quality of all TEE image sets (i.e. before and after suctioning) post hoc. The acquired numeric scales were combined, and compared before and after suctioning, and calculated how much percentage of patients had improved image quality (i.e. increase in numeric scale), same quality (i.e. same numeric scale), and worsened image quality (i.e. decrease in numeric scale)
Time Frame: TEE image sets were acquired after general anesthesia induction (before suction) and after 10minutes (after suction), and the outcome was the difference in image quality. In 6-8 months, investigator C did the same analysis on the same images in one day.
Population: Surgeries which need intraoperative TEE (cardiac or liver transplant surgery)
Measure: Count of Units; unit: image sets
Units Other Than Participants: image sets
Groups:
- TEE Image Before and After Suction: Suction orogastric tube which is attached to TEE probe
Arm/Group | TEE Image Before and After Suction
Number analyzed (Participants) | 47
Number analyzed (image sets) | 141
image sets
  Improved after suction | 79
  Same after suction | 62
  Worse after suction | 0

2. Secondary Outcome: Reproducibility of the Left Ventricular Fraction Area Change (LV FAC) (Inter-observer)
Description: The reproducibility of the LV FAC was assessed, assuming that better image quality would yield better LV FAC reproducibility. Three investigators (A, B, and C) assessed the quality of tall TEE image sets (i.e. before and after suction) post oc. These image sets were combined, and assessment was done for each group (i.e. before and after suctioning)
Time Frame: Images are acquired after general anesthesia induction (before suctioning) and after 10min (after suctioning)
Population: Patients who need intraop TEE for cardiac surgery and liver transplant surgery)
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient
Units Other Than Participants: image sets
Arm/Group | TEE Image Before and After Suction
Number analyzed (Participants) | 47
Number analyzed (image sets) | 141
intraclass correlation coefficient
  intraclass correlation coefficients of LV FAC before suction | 0.659 [0.511 to 0.78]
  intraclass correlation coefficients of LV FAC after suction | 0.903 [0.849 to 0.941]

3. Secondary Outcome: Reproducibility of the Left Ventricular Fraction Area Change (LV FAC) (Intra-observer)
Description: Investigator C assess all the image sets in one day again after 6-8 months to determine if there is intra-observer variability with the initial assessment of image quality, All investigators are blinded to which images are obtained before or after suction
Time Frame: 6-8 months after initial images obtained during surgery
Population: Patients who need intraop TEE for cardiac surgery and liver transplant surgery)
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient
Units Other Than Participants: image sets
Arm/Group | TEE Image Before and After Suction
Number analyzed (Participants) | 47
Number analyzed (image sets) | 47
intraclass correlation coefficient
  intraclass correlation coefficients of LV FAC before suction | 0.716 [0.536 to 0.833]
  intraclass correlation coefficients of LV FAC after suction | 0.935 [0.887 to 0.963]

ADVERSE EVENTS:
Time Frame: 1 month
Description: Esophageal trauma, stomach trauma, GI bleed, dysphagia, or anything related to TEE
Groups:
- TEE Related Complications: Esophageal trauma, stomach trauma, GI bleed, dysphagia
Arm/Group | TEE Related Complications
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT03454399/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT03454399/ICF_001.pdf